CLINICAL TRIAL: NCT04543383
Title: A Two-Part, Open-Label, Randomized, Placebo-Controlled Crossover Study to Assess the Reversal of the Anticoagulant Effects of Milvexian by 4-Factor Prothrombin Complex Concentrate (4F-PCC) (Part 1) and Recombinant Human Factor VIIa (rFVIIa) (Part 2) in Healthy Subjects
Brief Title: A Study to Assess the Reversal of the Anticoagulant Effects of Milvexian by 4-Factor Prothrombin Complex Concentrate (4F-PCC) (Part 1) and Recombinant Human Factor VIIa (rFVIIa) (Part 2) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108769; 2020-000180-24 (EudraCT Number); 70033093EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-07-28; First posted 2020-09-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — milvexian; Factor IX; recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Participants will receive two oral doses of milvexian (on Days 1 to 3), one in the morning and one in the evening. On Day 4, participants will only receive the morning dose of milvexian. On Day 4, four hours after the morning dosing of milvexian, each participant will receive an intravenous (IV) infusion of 4-Factor Prothrombin Complex Concentrate (4F-PCC) or matching placebo as per the treatment sequence AB and BA; in treatment period 1 and treatment period 2 where Treatment A=Dose 2 of milvexian + Dose 1 of 4F-PCC; Treatment B=Dose 2 milvexian + Placebo. A washout period of 14 days to 21 days will be maintained between each treatment period 1 and 2.
  Interventions: Drug: Milvexian; Biological: 4-Factor Prothrombin Complex Concentrate (4F-PCC); Biological: Placebo matching to 4F-PCC
- Part 2 (Group 1) (Experimental): Participants will receive an oral dose of milvexian in morning in fed state on Day 1 and IV injection of Recombinant Human Factor VIIa (rFVIIa) or placebo matching to rFVIIa on Day 1 after 4 hours post morning milvexian dose in the following treatment sequence: DEF1, EF1D, F1DE, EDF1, F1ED and DF1E; in treatment period 1, treatment period 2 and treatment period 3 respectively where Treatment D=Dose 1 of milvexian +Dose 1 of rFVIIa; Treatment E=Dose 3 of milvexian+Dose 1 of rFVIIa; Treatment F1=Dose 3 of milvexian+Placebo; Treatment F2=Dose 1 of milvexian+Placebo. A washout period of 4 days will be maintained between each treatment period 1, 2 and 3.
  Interventions: Drug: Milvexian; Biological: Recombinant Human Factor VIIa (rFVIIa); Biological: Placebo matching to rFVIIa
- Part 2 (Group 2) (Experimental): Participants will receive an oral dose of milvexian in morning in fed state on Day 1 and IV injection of rFVIIa or placebo matching to rFVIIa on Day 1 after 4 hours post morning milvexian dose in the following treatment sequence: DEF2, EF2D, F2DE, EDF2, F2ED and DF2E; in treatment period 1, treatment period 2 and treatment period 3 respectively where Treatment D=Dose 1 of milvexian+Dose 1 of rFVIIa; Treatment E=Dose 3 of milvexian+Dose 1 of rFVIIa; Treatment F1=Dose 3 of milvexian+Placebo; Treatment F2=Dose 1 of milvexian+Placebo. A washout period of 4 days will be maintained between each treatment period 1, 2 and 3.
  Interventions: Drug: Milvexian; Biological: Recombinant Human Factor VIIa (rFVIIa); Biological: Placebo matching to rFVIIa

INTERVENTIONS:
Drug: Milvexian — Milvexian will be administered orally.
  Other Names: BMS-986177; JNJ-70033093
Biological: 4-Factor Prothrombin Complex Concentrate (4F-PCC) — 4F-PCC will be administered intravenously.
  Arms: Part 1
Biological: Recombinant Human Factor VIIa (rFVIIa) — rFVIIa will be administered intravenously.
  Arms: Part 2 (Group 1); Part 2 (Group 2)
Biological: Placebo matching to 4F-PCC — Placebo matching to 4F-PCC will be administered intravenously.
  Arms: Part 1
Biological: Placebo matching to rFVIIa — Placebo matching to rFVIIa will be administered intravenously.
  Arms: Part 2 (Group 1); Part 2 (Group 2)

SUMMARY:
The primary purpose of this study is to evaluate the reversal of the anticoagulant effects of milvexian by 4-Factor Prothrombin Complex Concentrate (4F-PCC) and Recombinant Human Factor VIIa (rFVIIa) in healthy participants as measured by changes from baselines of the coagulation testing parameters (activated partial thromboplastin time [aPTT] and thrombin generation assay [TGA]).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy on the basis of medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory test results, including serum chemistry, lipid profiles (low-density lipoprotein [LDL], high-density lipoprotein [HDL], apolipoprotein B and lipoprotein a), levels of protein C, protein S and antithrombin, fibrinogen, factors VIIIc, IXc, Xc, XIc and blood coagulation (activated partial thromboplastin time [aPTT], prothrombin time [PT]) measured at local laboratory, hematology and urinalysis performed at screening. If abnormalities or deviations from normal are observed, they must be of no clinical significance in the opinion of the investigator
* Before randomization, a woman must either be: Not of childbearing potential defined as: Postmenopausal-A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level greater than (>) 40 International Units Per Liter (IU/L) or milli-international units per milliliter (mIU/mL) in the postmenopausal range may be used to confirm a postmenopausal state in women, however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient; Permanently sterile- Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Of childbearing potential, a woman must have an intrauterine device without estrogen- and or progestogen-containing system, or have vasectomized partner or practice sexual abstinence, agrees to remain on the above highly effective contraceptive method throughout the study and for at least 90 days after the last dose of study intervention
* A male participant must wear a condom when engaging in any activity with a woman of childbearing potential during the study and for the duration of treatment with milvexian plus 5 half-lives of the study intervention for a total of 94 days after the completion of treatment. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception because condom may break or leak
* If a woman, must have a negative highly sensitive serum (Beta-human chorionic gonadotropin [Beta-hCG]) pregnancy test at screening and urine (Beta-hCG) pregnancy test on Day -1 of each study period (Part 1) or on Day -1 of Period 1 (Part 2)
* Women must have no history of excessive menstrual bleeding or hemorrhage following pregnancy delivery
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for 94 days after receiving the last dose of study intervention
* Body mass index (weight [kilogram {kg}/height^2 [meter {m^2}]) more than equal to 18.0 and less than equal to 29.9 kg/m^2 body weight not less than 50 kg and not more than 100 kg.

Exclusion Criteria:

* History or family history of any known illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study intervention to the participant or that could prevent, limit or confound the protocol specified assessments. This may include but is not limited to any known bleeding or clotting disorder, cardiolipin antibody and anti-beta2-glycoprotein I, abnormal levels of fibrinogen, factors VIIIc, IXc, Xc, XIc, inherited or acquired thrombophilia, bleeding diathesis or coagulopathy, excessive bruising, bleeding from nose or gums or known disorders with increased bleeding risk, serious bleeding including gastrointestinal bleeding requiring hospitalization, intracranial bleeding of any type, or uncontrollable postoperative bleeding, a history of arterial or venous thrombosis, phlebitis, inherited or acquired thrombophilia, known family history of unexplained thrombotic disorders, known intracranial or intraabdominal tumor, hemorrhage, or aneurysm, liver or renal dysfunction, clinically significant cardiac, vascular disorders, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic abnormalities, or metabolic disturbances, or poor venous access
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders criteria within 1 year before screening or positive test result(s) for alcohol and/or drugs of abuse (such as hallucinogens (lysergic acid diethylamide [LSD]), barbiturates, opiates, opioids, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening and/or on Day -1 of Period 1
* Have laboratory values at screening or Day -1 of Period 1 above or below limits of normal that in the investigator's judgment may affect the safety of the participants
* Any of the following laboratory results outside of the ranges specified below at screening or on Day -1 of Period 1, confirmed by repeat: Hemoglobin or hematocrit < lower limit of normal, Platelet count less than (<) lower limit of normal, aPTT, or PT > upper limit of normal (ULN), LDL, HDL, apolipoprotein B, or lipoprotein a, outside the normal reference ranges, Factor II gene mutation or Factor V Leiden mutation assessed by polymerase chain reaction (PCR) tests, positive for Lupus Anticoagulants (LA screen, confirm and Silica Clotting Time [SCT]), cardiolipin antibody and anti-beta2-glycoprotein I, abnormal levels of protein C, protein S, antithrombin, fibrinogen, factors VIIIc, IXc, Xc, XIc
* Any of the following on 12-lead ECG based on an average of triplicate measurements at screening or Day -1 of Period 1: PR greater than or equal to (>=) 210 millisecond (msec), QRS >=120 msec, QTcF>=450 msec for male and >=470 msec for female, Heart Rate (HR) >= 100 beats per minute (bpm)
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) and known allergy to the study interventions or any of the excipients of the formulations. History of allergy to or unwillingness to consume any component of high-fat breakfast menu to be provided in this study

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Change from Baseline in Activated Partial Thromboplastin Time (aPTT) | Baseline, Day 4
  The aPTT measures the time it takes plasma to clot when exposed to substances that activate the contact factors, which assesses the intrinsic and common pathways of coagulation.
Part 2: Change from Baseline in aPTT | Baseline, Day 1
  The aPTT measures the time it takes plasma to clot when exposed to substances that activate the contact factors, which assesses the intrinsic and common pathways of coagulation.
Part 1: Change from Baseline in Endogenous Thrombin Potential (ETP) (Thrombin Generation Assay [TGA] Parameter) | Baseline, Day 4
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the ETP (TGA parameter). The ETP assesses the amount of thrombin which can be generated after the in vitro activation of coagulation and represents the balance between pro and anti-coagulant forces in plasma.
Part 1: Change from Baseline in Lag Time (TGA Parameter) | Baseline, Day 4
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the lag time (TGA parameter). The lag time is defined as the time needed until thrombin is generated.
Part 1: Change from Baseline in Peak Thrombin (TGA Parameter) | Baseline, Day 4
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the peak thrombin (TGA parameter). The peak thrombin is defined as the maximal effect on thrombin generation.
Part 1: Change from Baseline in Time to Peak Thrombin (TGA Parameter) | Baseline, Day 4
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the time to peak thrombin (TGA parameter). The time to peak thrombin is defined as the time required to reach maximal effect on thrombin generation.
Part 2: Change from Baseline in ETP (TGA Parameter) | Baseline, Day 1
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the ETP (TGA parameter). The ETP assesses the amount of thrombin which can be generated after the in vitro activation of coagulation and represents the balance between pro and anti-coagulant forces in plasma.
Part 2: Change from Baseline in Lag Time (TGA Parameter) | Baseline, Day 1
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the lag time (TGA parameter). The lag time is defined as the time needed until thrombin is generated.
Part 2: Change from Baseline in Peak Thrombin (TGA Parameter) | Baseline, Day 1
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the peak thrombin (TGA parameter). The peak thrombin is defined as the maximal effect on thrombin generation.
Part 2: Change from Baseline in Time to Peak Thrombin (TGA Parameter) | Baseline, Day 1
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the time to peak thrombin (TGA parameter). The time to peak thrombin is defined as the time required to reach maximal effect on thrombin generation.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAE) as a Measure of Safety and Tolerability | Part 1: Up to 74 Days; Part 2: Up to 25 Days
  Treatment-emergent adverse events (TEAEs) are defined as adverse events (AEs) with onset or worsening on or after date of first dose of study treatment.
Number of Participants with TEAEs of interest | Part 1: Up to 74 Days; Part 2: Up to 25 Days
  Number of participants with TEAEs of interest will be reported. TEAEs associated with the following situations are considered as TEAEs of interest: bleeding, thromboembolic events (TEs) and liver injury.
Parts 1 and 2: Change From Baseline in Pulse Rate | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Changes from baseline in pulse rate will be assessed.
Parts 1 and 2: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Changes from baseline in SBP and DBP will be assessed.
Parts 1 and 2: Change From Baseline in QTc Interval | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by ECG.
Parts 1 and 2: Change from Baseline in Heart Rate (HR) | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in HR will be measured by ECG.
Parts 1 and 2: Change from Baseline in QRS Interval | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in QRS interval will be measured by ECG
Parts 1 and 2: Change from Baseline in PR Interval | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in PR interval will be measured by ECG.
Parts 1 and 2: Change From Baseline in QT Interval | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in QT interval will be measured by ECG.
Parts 1 and 2: Change From Baseline in Hematology Parameter: Platelet Count | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameter (platelet count) will be assessed.
Parts 1 and 2: Change From Baseline in Hematology Parameter: Red Blood Cell (RBC) count | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameter (RBC count [Unit: Cells per liter]) will be assessed.
Parts 1 and 2: Change From Baseline in Hematology Parameter: Hemoglobin (Hb) | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameter (Hb [Grams per deciliter]) will be assessed.
Parts 1 and 2: Change From Baseline in Hematology Parameter: Hematocrit | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameter (Hematocrit) will be assessed.
Parts 1 and 2: Change From Baseline in Hematology Parameter: Mean Corpuscular Volume (MCV) | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameter (MCV [Femtoliter]) will be assessed.
Parts 1 and 2: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin (MCH) | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameter (MCH [Picogram]) will be assessed.
Parts 1 and 2: Change From Baseline in Hematology Parameter: Percentage of Reticulocytes | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameter (Percentage of reticulocytes) will be assessed.
Parts 1 and 2: Change From Baseline in Hematology Parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in hematology parameters (Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils [Unit: Giga cells per liter]) will be assessed.
Parts 1 and 2: Change From Baseline in Coagulation Parameter: Activated Partial Thromboplastin Time (aPTT) and Prothrombin Time (PT) | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in coagulation parameter (aPTT and PT [Unit: Seconds]) will be assessed.
Parts 1 and 2: Change from Baseline in Serum Chemistry Parameters: Bicarbonate, Calcium, Glucose, Chloride, Magnesium, Phosphate, Sodium, BUN, Cholesterol, HDL, LDL, Triglycerides | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in serum chemistry parameters (Bicarbonate, Calcium, Glucose, Chloride, Magnesium, Phosphate, Sodium, Blood urea nitrogen [BUN], Cholesterol, High density Lipoprotein [HDL], Low density lipoprotein [LDL], Triglycerides [Unit: Millimole per Liter]) will be assessed.
Parts 1 and 2: Change from Baseline in Serum Chemistry Parameters: ALT, AST, GGT, LDH, Alkaline phosphatase, CPK | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in serum chemistry parameters (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], Gamma-glutamyl transferase [GGT], Lactic acid dehydrogenase [LDH], Alkaline phosphatase, Creatine phosphokinase [CPK] [Unit: International units per Liter]) will be assessed.
Parts 1 and 2: Change from Baseline in Serum Chemistry Parameters: Amylase | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in serum chemistry parameters (Amylase [Unit: Units per liter]) will be assessed.
Parts 1 and 2: Change from Baseline in Serum Chemistry Parameters: Lipase | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in serum chemistry parameters (Lipase [Unit: Units per liter]) will be assessed.
Parts 1 and 2: Change from Baseline in Serum Chemistry Parameters: Total Bilirubin, Creatinine and Uric Acid | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in serum chemistry parameters (Total bilirubin, Creatinine and Uric acid [Unit: Micromoles per Liter]) will be assessed.
Parts 1 and 2: Change from Baseline in Serum Chemistry Parameters: Total Protein and Albumin | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in serum chemistry parameters (Total protein and Albumin [Unit: Gram per Liter]) will be assessed.
Parts 1 and 2: Change From Baseline in Urinalysis Parameter: Specific Gravity | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in urinalysis parameter (Specific gravity) tests will be assessed.
Parts 1 and 2: Change From Baseline in Urinalysis Parameter: pH | Part 1: Up to 77 Days; Part 2: Up to 59 Days
  Change from baseline in urinalysis parameter (pH) tests will be assessed.
Part 1: Mean Trough Plasma Concentration of Milvexian at Steady State (Ctrough) | Part 1: Predose, 2, 4, 4.75, 5, 6, 8, 12, 24, 48, and 72 hours Postdose
  Mean trough plasma concentration of milvexian at steady state will be reported.
Part 1 and Part 2: Maximum Observed Analyte Concentration (Cmax) of Milvexian | Part 1: Predose, 2, 4, 4.75, 5, 6, 8, 12, 24, 48, and 72 hours Postdose; Part 2: 0.25, 2, 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Cmax is the maximum observed analyte concentration.
Part 1 and Part 2: Time to Reach Maximum Plasma Concentration (Tmax) of milvexian | Part 1: Predose, 2, 4, 4.75, 5, 6, 8, 12, 24, 48, and 72 hours Postdose; Part 2: 0.25, 2, 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Tmax is defined as actual sampling time to reach the maximum observed analyte concentration.
Parts 1 and Part 2: Elimination Half-Life (t1/2) of Milvexian | Part 1: Predose, 2, 4, 4.75, 5, 6, 8, 12, 24, 48, and 72 hours Postdose; Part 2: 0.25, 2, 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  t1/2 elimination half-life means time measured for the plasma concentration to decrease by 1 half to its original concentration of milvexian.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Dosing Interval (AUC [0-t]) of Milvexian | Part 1: Predose, 2, 4, 4.75, 5, 6, 8, 12, 24, 48, and 72 hours Postdose
  Area under the plasma concentration versus time curve from time zero to dosing interval of milvexian.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Milvexian | Part 2: 0.25, 2, 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Area under the plasma concentration versus time curve from time zero to infinity with extrapolation of the terminal phase of milvexian.
Part 1 and Part 2: Area Under Plasma Concentration From Time Zero to the Last Quantifiable Concentration (AUC [0-last]) of Milvexian | Part 1: Predose, 2, 4, 4.75, 5, 6, 8, 12, 24, 48, and 72 hours Postdose; Part 2: 0.25, 2, 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Area under the plasma concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration of milvexian will be assessed.
Part 2: Maximum Observed Analyte Concentration (Cmax) of rFVIIa | Part 2: 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Cmax is the maximum observed analyte concentration.
Part 2: Time to Reach Maximum Plasma Concentration (Tmax) of rFVIIa | Part 2: 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Tmax is defined as actual sampling time to reach the maximum observed analyte concentration.
Part 2: Elimination Half-Life (t1/2) of rFVIIa | Part 2: 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  t1/2 elimination half-life means time measured for the plasma concentration to decrease by 1 half to its original concentration of rFVIIa.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of rFVIIa | Part 2: 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Area under the plasma concentration versus time curve from time zero to infinity with extrapolation of the terminal phase of rFVIIa.
Part 2: Area Under Plasma Concentration From Time Zero to the Last Quantifiable Concentration (AUC [0-last]) of rFVIIa | Part 2: 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  Area under the plasma concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration of rFVIIa will be assessed.
Part 2: Systemic Clearance (CL) of rFVIIa | Part 2: 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose will be estimated by dividing the total administered dose by the area under the plasma concentration-time curve from time zero to infinite time (AUC [0-infinity]).
Part 2: Volume of distribution (Vz) of rFVIIa | Part 2: 4, 4.25, 4.5, 5, 6, 8, 12, 24 hours Postdose
  The Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Part 1 and Part 2: Change from Baseline in aPTT | Part 1: Baseline, Day 1, Day 4, Day 5, Day 6 and Day 7; Part 2: Baseline, Day 1 and Day 2
  Change from baseline in aPTT will be reported.
Part 1 and Part 2: Change from Baseline in ETP (TGA Parameter) | Part 1: Baseline, Day 1, Day 4, Day 5, Day 6 and Day 7; Part 2: Baseline, Day 1 and Day 2
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the ETP (TGA parameter). The ETP assesses the amount of thrombin which can be generated after the in vitro activation of coagulation and represents the balance between pro and anti-coagulant forces in plasma.
Part 1 and Part 2: Change from Baseline in Lag Time (TGA Parameter) | Part 1: Baseline, Day 1, Day 4, Day 5, Day 6 and Day 7; Part 2: Baseline, Day 1 and Day 2
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the lag time (TGA parameter). The lag time is defined as the time needed until thrombin is generated.
Part 1 and Part 2: Change from Baseline in Peak Thrombin (TGA Parameter) | Part 1: Baseline, Day 1, Day 4, Day 5, Day 6 and Day 7; Part 2: Baseline, Day 1 and Day 2
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the peak thrombin (TGA parameter). The peak thrombin is defined as the maximal effect on thrombin generation.
Part 1 and Part 2: Change from Baseline in Time to Peak Thrombin (TGA Parameter) | Part 1: Baseline, Day 1, Day 4, Day 5, Day 6 and Day 7; Part 2: Baseline, Day 1 and Day 2
  The TGA measures the thrombin generation that is indicative of an overall coagulating capacity. A calibrated automated thrombography is used to monitor the concentration of thrombin in clotting plasma with a fluorogenic substrate. The data derived from the thrombography can be used to determine the time to peak thrombin (TGA parameter). The time to peak thrombin is defined as the time required to reach maximal effect on thrombin generation.
Percent Change from Baselines in aPTT | Part 1: Baseline, Day 1, Day 4, Day 5, Day 6 and Day 7; Part 2: Baseline, Day 1 and Day 2
  Percent change from baseline in aPTT will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency